CLINICAL TRIAL: NCT03297346
Title: Early Detection of Cardiovascular Changes After Radiotherapy for Breast Cancer (EARLY HEART Study) in the Frame of the Implications of MEDIcal Low Dose RADiation Exposure (MEDIRAD) European Project
Brief Title: Early Detection of Cardiovascular Changes After Radiotherapy for Breast Cancer
Acronym: EARLY-HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Radioprotection et de Surete Nucleaire (Other Government)
Collaborators: Academisch Ziekenhuis Groningen (Other); Technical University of Munich (Other); Institut Català d'Oncologia (Other); Hospital de Santa Maria, Portugal (Other); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Principal Investigator, Sophie JACOB, PhD, Institut de Radioprotection et de Surete Nucleaire
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MEDIRAD EARLY-HEART_1.2
Record Dates: First submitted 2017-09-21; First posted 2017-09-29 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer Female
Keywords: radiotherapy; cardiovascular changes; cardiac imaging; circulating biomarkers; dosimetry

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer patients treated with RT (Other): Cardiac imaging and circulating biomarkers measurements to evaluate:
  * myocardial dysfunction and deformation (ECHO-ST)
  * coronary artery lesions and coronary artery calcium score (CT)
  * myocardium including tissue abnormalities, cardiac morphology and function (MRI)
  * blood-based biomarkers of cardiovascular changes (BLOOD)
  Interventions: Other: Cardiac imaging and circulating biomarkers

INTERVENTIONS:
Other: Cardiac imaging and circulating biomarkers — Automated 2D-speckle-tracking echocardiography (ECHO-ST); Computed tomography coronary angiography (CT); Cardiac magnetic resonance imaging (MRI); Blood samples for circulating biomarkers measurements (BLOOD)

SUMMARY:
Breast cancer (BC) radiotherapy leads to coincidental radiation of the heart, resulting in increased risk of a variety of heart diseases. Identifying BC patients with the highest risk of radiation-induced cardiac complications is crucial for developing strategies for primary and secondary prevention. Little has been done on the relationship between dose distribution to different anatomical cardiac structures during radiotherapy and early cardiovascular changes that may lead to cardiac complications.

In the framework of the European project MEDIRAD, the EARLY-HEART multicenter prospective cohort was launched in August 2017, involving 5 investigating centers from France, Netherlands, Germany, Spain and Portugal. With 250 BC patients prospectively followed for 2 years, the main objective is to identify and validate the most important cardiac imaging (echocardiography, computed tomography coronary angiography, cardiac magnetic resonance imaging) and circulating biomarkers of radiation-induced cardiovascular changes arising in the first 2 years after BC radiotherapy.

DETAILED DESCRIPTION:
EARLY-HEART is a multicentre prospective cohort study that will include 250 female primary breast cancer cases aged 40-75 years treated with postoperative radiotherapy (RT) alone after breast-conserving surgery using modern planning-CT based RT technologies and followed for 2 years after RT in one of the 5 participating hospitals. In addition to the standard follow-up, patients will need to give repeated blood samples and will undergo repeated cardiac imaging:

* Functional and anatomical cardiac imaging biomarkers will be based on automated 2D-speckle-tracking echocardiography (ECHO-ST); Computed Tomography Coronary Angiography (CT) and cardiac magnetic resonance imaging (MRI).
* Circulating biomarkers (BLOOD) will be based on a panel of multiple classical or novel blood-based biomarkers.

Imaging and circulating biomarkers measurements will be assessed at baseline before RT (ECHO, CT, MRI, BLOOD); at the end of RT (BLOOD); 6 months after RT (ECHO, MRI, BLOOD) and 24 months after RT (ECHO, CT, MRI, BLOOD).

Changes in functional and anatomical cardiac imaging and circulating biomarkers between unexposed status before RT and exposed status after RT at different time points will be first analysed to evaluate the effects of RT on the heart.

All relevant DICOM-data (including planning-CT scans and the ECHO, MRI and CT) will be centralized to the MEDIRAD-ENACT database managed by University of Groningen for automated segmentation of all cardiac substructures (including coronary arteries) to ensure uniformity of the segmentation procedure between centres. The RT planning CTs will be used to generate dose volume histograms and 3D dose maps of the heart and cardiac substructures in order to correlate the localization of any cardiovascular change with the anatomical dose distribution.

In the presence of a cardiac outcome, a multimetric Normal Tissue Complication Probability (NTCP) individual risk model will be constructed and an integrative clinical-biologic risk score will be developed for individual risk prediction.

ELIGIBILITY:
Inclusion Criteria:

* Female unilateral breast cancer patients
* Treated with primary breast conserving surgery for stage I-III invasive adenocarcinoma of the breast or ductal carcinoma in situ (DCIS)
* Age between 40-75 years at time of start radiotherapy
* World Health Organisation (WHO) performance status 0-1
* Planned for radiotherapy alone to the breast with or without the lymph node areas
* Radiotherapy based on planning-CT scan using either three dimensional conformal radiation therapy (3D-CRT), Intensity-modulated radiotherapy (IMRT), or Volumetric Arc Therapy (VMAT/RapidArc)
* Written Informed consent

Exclusion Criteria:

* Male breast cancer patients
* Neoadjuvant or adjuvant chemotherapy
* M1 disease (metastatic breast cancer)
* Medical history of coronary artery disease and/or myocardial infarction and/or atrial fibrillation
* Previous thoracic or mediastinal radiation
* Contraindications to injection of iodinated contrast such as allergy or renal failure
* Pregnancy or lactation
* Atrial fibrillation detected during electrocardiogram before radiotherapy
* Abnormal echocardiography before radiotherapy defined as: Left Ventricular Ejection Fraction<50%; longitudinal strain ≤ -16%; longitudinal strain rate <-1%, and/or abnormal wall motion
* Presence of myocardial infarction detected during MRI before radiotherapy
* CT or MRI results before radiotherapy requiring revascularisation

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with decreased myocardial function assessed by echocardiography | 2 years after radiotherapy (baseline measurements performed before radiotherapy)
  Number of patients with an increased of at least 2.5% in the Global Longitudinal Strain (GLS) between baseline and 2 years after radiotherapy

SECONDARY OUTCOMES:
Changes in myocardial function measurements assessed by echocardiography | 6 months and 2 years after radiotherapy (baseline measurements performed before radiotherapy)
  Increase of the segmental strain measurements (unit of measures:%)
Anatomical changes in coronary arteries assessed by cardiac CT | 2 years after radiotherapy (baseline measurements performed before radiotherapy)
  Increase of the number of coronary segments containing any plaque or increase of the calcium score
Myocardial tissue abnormalities assessed by cardiac MRI | 6 months and 2 years after radiotherapy (baseline measurements performed before radiotherapy)
  Increase of the native mean myocardial T1 mapping value
Changes in circulating biomarkers measurements | at the end of radiotherapy (through radiotherapy completion, an average of 5 weeks after starting date of radiotherapy), 6 months and 2 years after radiotherapy (baseline measurements performed before radiotherapy)
  Significant increase or decrease in the following biomarkers:
  classical biomarkers of cardiac injury (C-reactive protein, Troponin I, Troponin T, B-type natriuretic peptide (BNP), N-terminal pro-brain natriuretic peptide (NT-Pro BNP), beta2-Microglobulin, Galectin 3); Inflammatory cytokines; biomarkers of endothelial activation and dysfunction; Microparticles; MicroRNAs; circulating DNA methylation

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Jacob, PhD, Study Chair — Institut de Radioprotection et de Sûreté Nucléaire
Locations (5):
- IRSN - Clinique Pasteur, Toulouse, France
- Klinikum rechts der Isar der Technischen Universität München, Munich, Germany
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Associação para Investigação e Desenvolvimento da Faculdade de Medicina, Lisbon, Portugal
- Institut Català d'Oncologia, Girona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Locquet M, Spoor D, Crijns A, van der Harst P, Eraso A, Guedea F, Fiuza M, Santos SCR, Combs S, Borm K, Mousseaux E, Gencer U, Frija G, Cardis E, Langendijk H, Jacob S. Subclinical Left Ventricular Dysfunction Detected by Speckle-Tracking Echocardiography in Breast Cancer Patients Treated With Radiation Therapy: A Six-Month Follow-Up Analysis (MEDIRAD EARLY-HEART study). Front Oncol. 2022 Jun 28;12:883679. doi: 10.3389/fonc.2022.883679. eCollection 2022. PMID 35837099
- [Derived] Walker V, Crijns A, Langendijk J, Spoor D, Vliegenthart R, Combs SE, Mayinger M, Eraso A, Guedea F, Fiuza M, Constantino S, Tamarat R, Laurier D, Ferrieres J, Mousseaux E, Cardis E, Jacob S. Early Detection of Cardiovascular Changes After Radiotherapy for Breast Cancer: Protocol for a European Multicenter Prospective Cohort Study (MEDIRAD EARLY HEART Study). JMIR Res Protoc. 2018 Oct 1;7(10):e178. doi: 10.2196/resprot.9906. PMID 30274965

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT03297346/Prot_SAP_ICF_000.pdf